CLINICAL TRIAL: NCT00087048
Title: The Use Of Weekly Topotecan As Second Line Therapy In Small Cell Lung Cancer
Brief Title: Topotecan in Treating Patients With Recurrent Extensive-Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000372872; CASE-HFHS-1503; HFH-HFHS-1503; HFH-HFHS-0205; CWRU-050308
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well high-dose topotecan works as second-line therapy in treating patients with recurrent extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall survival of patients with recurrent extensive stage small cell lung cancer treated with high-dose topotecan hydrochloride.

Secondary

* Determine the safety and toxic effects of this drug in these patients.
* Determine the recurrence-free survival of patients treated with this drug.
* Determine time to response and tumor response in patients treated with this drug.
* Determine the quality of life of patients treated with this drug.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive high-dose topotecan hydrochloride IV over 30 minutes on days 1, 8, 15, 22, 29, and 36. Treatment repeats every 56 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, day 1 of each course (except course 1), at the end of study treatment, and then every 3 months thereafter.

Patients are followed at 7-14 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed small cell lung cancer (SCLC)

  * Recurrent extensive stage disease
  * No mixed histology
* Measurable disease

  * At least 1 bidimensionally measurable, non-central nervous system (CNS), indicator lesion confirmed by CT scan or MRI
* Sensitive disease

  * Responded to prior first-line therapy AND relapsed ≥ 60 days after response (90 days after initiation of first-line therapy)
* Eligible for high-dose chemotherapy
* No symptomatic brain metastases affecting performance status

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-2

Life expectancy

* At least 2 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Hematocrit > 35% (without transfusion)

Hepatic

* Serum glutamic-oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) ≤ 2 times normal*
* Alkaline phosphatase ≤ 2 times normal*
* Bilirubin ≤ 2.0 mg/dL
* Albumin > 2.5 g/dL
* Hepatitis B surface antigen negative
* No significant hepatic disease Note: *≤ 5 times upper limit of normal if liver metastases are present

Renal

* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* No history of cardiac arrhythmias
* No congestive heart failure
* No ischemic heart disease
* No stroke or other embolic disease requiring daily treatment that would preclude study participation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* HIV negative
* No known seizure disorder
* No active infection requiring systemic therapy within the past 2 weeks
* No known hypersensitivity to topotecan hydrochloride
* No medical or psychiatric condition that would preclude study participation
* No other malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or stage A low-grade prostate cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 4 weeks since prior antineoplastic and/or myelosuppressive chemotherapy
* No more than 1 prior chemotherapy regimen (except for adjuvant chemotherapy) for SCLC
* No prior topotecan hydrochloride

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 2 months since prior investigational agent
* No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2004-04; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Safety and toxic effects
Recurrence-free survival
Time to response and tumor response
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, MD, Study Chair — Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Case Comprehensive Cancer Center, Cleveland, Ohio